CLINICAL TRIAL: NCT02022670
Title: Clinical Translation of Nitrite Therapy to Treat Arterial Aging in Humans
Brief Title: Sodium Nitrite to Treat Arterial Aging
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: TheraVasc Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21HL107105 (NIH)
Record Dates: First submitted 2013-12-13; First posted 2013-12-30 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Vascular Aging
Keywords: endothelial function; arterial stiffness; flow-mediated dilation; pulse wave velocity; sodium nitrite; aging; vascular diseases
MeSH Terms: conditions — Vascular Diseases | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): inert oral capsules (0 mg sodium nitrite morning; 0 mg sodium nitrite in evening) for 10 weeks
  Interventions: Drug: Placebo
- Sodium Nitrite 80 mg/d (Experimental): 80 mg/day (40 mg in morning; 40 mg in evening) oral capsules for 10 weeks
  Interventions: Drug: Sodium Nitrite
- Sodium Nitrite 160 mg/d (Experimental): 160 mg/day (80 mg in morning; 80 mg in evening) oral capsules for 10 weeks
  Interventions: Drug: Sodium Nitrite

INTERVENTIONS:
Drug: Placebo — Sugar pill manufactured to mimic sodium nitrite capsules
  Arms: Placebo
Drug: Sodium Nitrite — 80 mg/d or 160 mg/d
  Other Names: TV1001
  Arms: Sodium Nitrite 160 mg/d; Sodium Nitrite 80 mg/d

SUMMARY:
The proposed research will determine the effectiveness of nitrite, a naturally occurring compound in the body, for improving the health and function of arteries in middle-aged and older adults. The study also will provide insight into how sodium nitrite therapy improves artery health by determining the physiological mechanisms (biological reasons) involved. Overall, the proposed research will provide important new scientific evidence on the effectiveness of sodium nitrite for decreasing the risk of developing cardiovascular diseases with aging.

DETAILED DESCRIPTION:
The improvement in blood vessel function and stiffness will be determined over a 10 week period. Subjects will be randomly assigned to either placebo (0 mg/day), low dose (80 mg/day) or high dose (160 mg/day) sodium nitrite. Main outcome measures will be performed at baseline and week 10.

ELIGIBILITY:
Inclusion Criteria:

* 50-79 years of age
* Ability to provide informed consent
* Score greater than 22 on the mini mental state exam
* Blood pressure greater than 100/60 mmHg for past 3 months

Exclusion Criteria:

* Are taking any of the following medications/drugs: hormone replacement therapy, anti-hypertensives, nitrates, nervous system depressants, allopurinol, phosphodiesterase-5 inhibitors, blood thinners
* Are currently sick/have chronic clinical diseases such as kidney disease, diabetes, or unstable cardiovascular disease
* Are hypersensitive to nitrates or nitrites
* Have glucose-6-phosphate dehydrogenase deficiency
* Have blood methemoglobin greater than 2%
* Have a BMI greater than 40 kg/m^2
* Have a baseline FMD of greater than 6%
* Have not been post-menopausal for at least 1 year
* Perform regular vigorous aerobic/endurance exercise

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Seals, Ph.D., Principal Investigator — University of Colorado, Boulder; Allison E DeVan, Ph.D., Study Director — University of Colorado, Boulder
Locations (1):
- Clinical Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- See also: Integrative Physiology of Aging Laboratory Website — http://www.colorado.edu/intphys/research/cardiovascular.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy men and women ages 50-79 years free of overt cardiovascular or chronic diseases.
Period: Overall Study
Arm/Group | Placebo | Sodium Nitrite 80 mg/d | Sodium Nitrite 160 mg/d
Started | 11 | 10 | 12
Completed | 10 | 10 | 11
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sodium Nitrite 80 mg/d | Sodium Nitrite 160 mg/d | Total
Number analyzed (Participants) | 11 | 10 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 60 (6) | 64 (6) | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 16
  Male | 6 | 5 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Baseline and Week 10 Flow-Mediated Dilation
Description: Brachial artery flow mediated dilation (FMD) is assessed prior to entering the study. If subjects pass the inclusion requirements, FMD is analyzed at baseline and week 10. Flow-Mediated Dilation is calculated as the percent change in artery diameter in response to 5 minutes of cuff occlusion at Baseline and Week 10 timepoints; i.e. (Peak Diameter-Baseline Diameter)/Baseline Diameter x 100.
Time Frame: Baseline (Week 0), Week 10
Measure: Mean (Standard Error); unit: %Change
Arm/Group | Placebo | Sodium Nitrite 80 mg/d | Sodium Nitrite 160 mg/d
Number analyzed (Participants) | 10 | 10 | 10
%Change
  Baseline | 3.120 (0.528) | 4.307 (0.501) | 3.118 (0.483)
  Week 10 | 3.740 (0.509) | 6.833 (0.785) | 4.609 (0.720)

2. Secondary Outcome: Baseline and Week 10 Plasma Nitrite Concentrations
Time Frame: Baseline (Week 0), Week 10
Measure: Mean (Standard Error); unit: micromolar
Arm/Group | Placebo | Sodium Nitrite 80 mg/d | Sodium Nitrite 160 mg/d
Number analyzed (Participants) | 10 | 10 | 11
micromolar
  Baseline | 0.201 (0.066) | 0.209 (0.053) | 0.155 (0.044)
  Week 10 | 0.261 (0.051) | 0.412 (0.066) | 0.369 (0.064)

3. Secondary Outcome: Baseline and Week 10 Aortic Pulse Wave Velocity
Time Frame: Baseline (Week 0), Week 10
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Placebo | Sodium Nitrite 80 mg/d | Sodium Nitrite 160 mg/d
Number analyzed (Participants) | 9 | 10 | 10
cm/sec
  Baseline | 782 (35) | 780 (55) | 946 (62)
  Week 10 | 774 (36) | 845 (75) | 942 (77)

ADVERSE EVENTS:
Arm/Group | Placebo | Sodium Nitrite 80 mg/d | Sodium Nitrite 160 mg/d
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 2/11 | 4/10 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | Sodium Nitrite 80 mg/d (N=10) | Sodium Nitrite 160 mg/d (N=12)
headache (General disorders) | 1 | 0 | 3
nausea (General disorders) | 1 | 0 | 0
fatigue (General disorders) | 0 | 2 | 2
dizziness/light-headedness (General disorders) | 1 | 1 | 2
asymptomatic orthostatic hypotension (General disorders) | 1 | 1 | 1
dry mouth (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No